CLINICAL TRIAL: NCT06460896
Title: Analysis of the Influence of Gastric By-Pass on the Pharmacokinetics of Common Drugs
Acronym: ABSORGYP
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP230873
Record Dates: First submitted 2024-05-30; First posted 2024-06-14 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2024-05

CONDITIONS: Bypass Bariatric Surgery
Keywords: bypass bariatric surgery, metabolic syndrome
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients eligible for bypass bariatric surgery and treated for metabolic syndrome (Other): 6 samples will be taken on the same day (T0, i.e. just before taking the drug, then T30 minutes, T1h, T2h, T4h, T7h after taking the drug).
  Interventions: Other: pharmacokinetic study

INTERVENTIONS:
Other: pharmacokinetic study — Multicenter pharmacokinetic study of the bioavailability of four compounds in GBP patients: candesartan, amlodipine, metformin and rosuvastatin.

SUMMARY:
Lack of knowledge of digestive absorption of drugs used in metabolic syndrome (MS) before and after gastric by-pass (GBP) in obese patients. The main objective is to study the changes in apparent clearance of candesartan, amlodipine, metformin and rosuvastatin, used in the treatment of metabolic syndrome in obese patients, between the preoperative period and 1 and 6 months after the performance of a GBP.

DETAILED DESCRIPTION:
The aim of this study is to investigate the pharmacokinetics of some of the most frequently prescribed oral drugs in hospital and outpatient medicine, in patients undergoing GBP surgery for obesity associated with metabolic syndrome. Paradoxically, despite their frequency of use, very few data, contradictory data or no data at all characterize the molecules we wish to study.

The number of patients undergoing GBP surgery is growing rapidly, as their life expectancy reaches that of the general population once their weight has normalized. However, while weight loss induced by surgery can improve, and more rarely cure, the comorbidities associated with metabolic syndrome, the majority of patients will need to continue or modify their treatments.

It is therefore essential to know the pharmacokinetics of the antihypertensive, lipid-lowering and hypoglycemic drugs they will be taking throughout their lives, in order to adapt their dosage if necessary, or even to change therapeutic class if their absorption is insufficient after GBP.

Moreover, as some studies have shown, the pharmacokinetics of many molecules are likely to vary over time in these patients (19), probably as a result of weight loss itself, but also possibly due to adaptive phenomena in the digestive tract. Studying the pharmacokinetics of the molecules used in the usual treatment of metabolic syndrome in most obese patients should make it possible to: target the preferred sites of absorption in the digestive tract of the molecules studied, study the variations in absorption linked to GBP but also the pharmacokinetic changes linked to weight loss as a function of time. In fact, metabolic capacity may be both decreased and increased in obese patients compared to healthy subjects (20,21), so that drug clearance may both increase and decrease after weight normalization. It is therefore difficult to predict the pharmacokinetics of drugs immediately or long after GYP. The results obtained should make it possible to adapt treatment in these patients, both in terms of changing the dosage administered and in the choice of molecules.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patients having undergone a complete bariatric course, eligible for bariatric surgery after validation of the operative indication by a multidisciplinary RCP dedicated to obesity, in accordance with HAS criteria: morbid obesity with BMI > 40 kg/m2 or severe obesity with BMI >35Kg/m2
* Patients with a comorbidity linked to one of the elements of metabolic syndrome that can be improved by surgery: type 2 diabetes, hypertension, dyslipidemia.
* Patients treated pre-operatively for at least 2 weeks with one or more of the molecules designed to control metabolic syndrome and selected for our study:

  * Antihypertensive: amlodipine; candesartan,
  * Hypolipidemic: rosuvastatin
  * Hypoglycemic agent: metformin
* Patients scheduled for Y-shaped gastric bypass surgery
* Membership of a social security scheme

Exclusion Criteria:

* History of restrictive bariatric surgery (sleeve)
* History of renal or hepatocellular insufficiency
* Patient undergoing treatment or having stopped treatment within the last month with a drug that may alter the clearance of the molecules studied: enzyme inducer or inhibitor (boosted antiproteases, macrolides, azole antifungals, grapefruit juice, rifampicin, rifabutin, phenobarbital, phenytoin, St John's wort), probenecid, non-steroidal anti-inflammatory drugs, etc.
* Patients treated with a drug that may alter the bioavailability of associated drugs: antacids containing aluminium or magnesium hydroxide, gastric dressings, etc.
* Patients for whom it is impossible to give informed consent (language barrier)
* Patients taking part in another interventional clinical study
* Patients under legal protection (guardianship, curatorship)
* Pregnant or breast-feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2027-09 (Estimated); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The main objective is to study the changes in apparent clearance of candesartan, amlodipine, metformin and rosuvastatin, used in the treatment of metabolic syndrome in obese patients | preoperative and postoperative phases at 1 month after surgery
  Difference in apparent clearance of study drugs between preoperative and postoperative phases at 1 month after surgery

SECONDARY OUTCOMES:
Determine changes in apparent clearance at 6 months after gastric bypass surgery compared with the pre-operative phase | pre-operative phase and 1 and 6 months after surgery
  Difference in apparent clearance of the 4 drugs studied between preoperative and postoperative phases at 6 months after gastric bypass surgery
Explain changes in apparent clearance as a function of weight loss | pre-operative phase and 1 and 6 months after surgery
  Change in apparent clearance as a function of body weight loss, measured by bioelectrical impedancemetry
Explain changes in apparent clearance as a function of changes in the fat/lean mass ratio | pre-operative phase and 1 and 6 months after surgery
  Change in apparent clearance as a function of change in body fat/lean mass ratio, measured by bioelectrical impedancemetry
Determine changes in apparent volumes of distribution between the pre-operative phase and 1 and 6 months after surgery | pre-operative phase and 1 and 6 months after surgery
  Differences in apparent volume of distribution values between the pre-operative phase and 1 month, then 6 months after surgery
Explain changes in apparent volumes of distribution as a function of body weight loss | pre-operative phase and 1 and 6 months after surgery
  Change in apparent volume of distribution as a function of body weight loss
Explain changes in apparent volumes of distribution as changes in body fat | pre-operative phase and 1 and 6 months after surgery
  Change in apparent volume of distribution as change in body fat/lean body mass ratio
Based on the results obtained, recommend any necessary changes in dosage or therapeutic class for these molecules | pre-operative phase and 1 and 6 months after surgery
  Dosages calculated to achieve the AUCs calculated before and 6 months after surgery, as well as the AUCs described for non-obese patients, at 1 month and 6 months post-surgery

CONTACTS AND LOCATIONS:
Overall Officials: Andrea LAZZATI, Principal Investigator — Assistance Publique de Paris
Locations (1):
- Service de chirurgie digestive, bariatrique et endocrinienne, Bobigny, France